CLINICAL TRIAL: NCT01862861
Title: Relieving Vasomotor Symptoms Effectively With Bioidentical Hormone Replacement Therapy: The REVERT Study
Acronym: REVERT
Status: Completed | Type: Observational
Sponsor: Medimix Specialty Pharmacy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Medimix Pharm-02
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Menopause
Keywords: Bioidentical Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Peri or post-menopausal women.: Women with peri or post-menopausal vasomotor symptoms between 30 and 60 years of age.

SUMMARY:
Bioidentical Hormone Replacement Therapy (BHRT) to assess a change in the number of various menopausal symptoms such as hot flashes and night sweats in surgically or naturally induced peri or post-menopausal women.

DETAILED DESCRIPTION:
Participants will be receiving a customized bioidentical hormone regimen which may include a combination of estrogens, progesterone, and testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be women who are in surgically or naturally induced menopause or perimenopause, as determined by their physician.
* Participants must be starting a new regimen of bioidentical hormone replacement therapy.
* Participants must be expected to receive therapy for at least 12 weeks.
* Participants must be between 30 and 65 years of age.
* Participants must be able to provide sound written informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf.

Exclusion Criteria:

* Participants must not have prior hypersensitivity or adverse events to any of the components in the customized prescription.
* Participants must not be pregnant or breastfeeding women.
* Participants must not be managed outside the Medimix Specialty Pharmacy system with regard to their bioidentical hormone replacement therapy.
* Participants must not be using another bioidentical hormone at the time of enrollment.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peri-menopausal or post-menopausal women between the age of 30 and 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of bioidentical hormone replacement therapy in decreasing the severity of vasomotor symptoms. | 12 Week Study
  The reduction of severity of vasomotor symptoms will be evaluated by utilizing the Menopause Rating Scale (MRS) from baseline to the end of study at 12 weeks.

SECONDARY OUTCOMES:
To evaluate health-related quality of life (HrQol) | 12 Weeks
  The quality of life (HrQol) will be evaluated by utilizing the Women's Health Questionnaire (WHQ)at baseline and at end of study at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Epstein, PharmD, Study Chair — The Medimix Specialty Pharmacy, LLC
Locations (1):
- The Medimix Specialty Pharmacy, LLC, Jacksonville, Florida, United States

REFERENCES:
- [Background] Wepfer ST. The science behind hormone replacement therapy, part ! Int J Pharm Compd. 2001 Nov-Dec;5(6):462-4. No abstract available. PMID 23982041
- [Background] Holtorf K. The bioidentical hormone debate: are bioidentical hormones (estradiol, estriol, and progesterone) safer or more efficacious than commonly used synthetic versions in hormone replacement therapy? Postgrad Med. 2009 Jan;121(1):73-85. doi: 10.3810/pgm.2009.01.1949. PMID 19179815
- [Background] Lorentzen J. Hormone replacement therapy: part 1 - the evolution of hormone treatment. Int J Pharm Compd. 2001 Sep-Oct;5(5):336-8. No abstract available. PMID 23981968
- [Background] Ruiz AD, Daniels KR, Barner JC, Carson JJ, Frei CR. Effectiveness of compounded bioidentical hormone replacement therapy: an observational cohort study. BMC Womens Health. 2011 Jun 8;11:27. doi: 10.1186/1472-6874-11-27. PMID 21651797
- [Background] Thurston RC, Joffe H. Vasomotor symptoms and menopause: findings from the Study of Women's Health across the Nation. Obstet Gynecol Clin North Am. 2011 Sep;38(3):489-501. doi: 10.1016/j.ogc.2011.05.006. PMID 21961716
- [Background] Gold EB, Colvin A, Avis N, Bromberger J, Greendale GA, Powell L, Sternfeld B, Matthews K. Longitudinal analysis of the association between vasomotor symptoms and race/ethnicity across the menopausal transition: study of women's health across the nation. Am J Public Health. 2006 Jul;96(7):1226-35. doi: 10.2105/AJPH.2005.066936. Epub 2006 May 30. PMID 16735636
- [Background] Levin ER, Hammes SR.Chapter 40. Estrogens and Progestins. In: Chabner BA, Bruton LL, Knollman BC, eds. Goodman & Gilman's The Pharmacological Basis of Therapeutics. 12nd ed. New York: McGraw-Hill; 2011. http://www.accesspharmacy.com/content.aspx?aID=16673417. Accessed September 28, 2012
- [Background] Snyder PJ. Chapter41. Androgens. In: Chabner BA, Bruton LL, Knollman BC, eds. Goodman & Gillman's The Pharmacological Basis of Therapeutics. 12nd ed. New York: McGraw-Hill; 2011. http;//www.accesspharmacy.com/content.aspx?aID=16673856. Accessed September 28,2012.
- [Background] Maclennan AH, Broadbent JL, Lester S, Moore V. Oral oestrogen and combined oestrogen/progestogen therapy versus placebo for hot flushes. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD002978. doi: 10.1002/14651858.CD002978.pub2. PMID 15495039
- [Background] Heinemann LA, DoMinh T, Strelow F, Gerbsch S, Schnitker J, Schneider HP. The Menopause Rating Scale (MRS) as outcome measure for hormone treatment? A validation study. Health Qual Life Outcomes. 2004 Nov 22;2:67. doi: 10.1186/1477-7525-2-67. PMID 15555079
- [Background] Hunter MS, The Women's Health Questionnaire (WHQ): the development, standardization and application of a measure of mid-aged women's emotional and physical health. Quality of Life Res. 2000;9(1):733-738.
- [Background] Clinical Pharmacology [database online]. Tampa, FL: Gold Standard, Inc.; 2012.
- [Background] Julious SA, Campbell MJ. Sample size calculations for paired or matched ordinal data. Stat Med. 1998 Jul 30;17(14):1635-42. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-k. PMID 9699235
- [Background] Julious SA, Campbell MJ, Altman DG. Estimating sample sizes for continuous, binary, and ordinal outcomes in paired comparisons: practical hints. J Biopharm Stat. 1999 May;9(2):241-51. doi: 10.1081/BIP-100101174. PMID 10379691